CLINICAL TRIAL: NCT06322095
Title: An Open Exploratory Study to Evaluate The Preliminary Efficacy of GH21 Combined With Primary Targeting or Immunotherapy in Patients With Advanced Solid Tumors Which Targeted or Immunotherapy Has Progressed
Brief Title: A Study of GH21 Combined With Previous Target Therapy or Immunotherapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH21C202
Record Dates: First submitted 2024-03-12; First posted 2024-03-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-03

CONDITIONS: Patients With Advanced Solid Tumor; Advanced Solid Tumor With Oncogenic Driver Mutations
MeSH Terms: interventions — 1,1'-(4,4'-(((5-chloropyrimidine-2,4-diyl)bis(azanediyl))bis(3-methoxy-4,1-phenylene))bis(piperazine-4,1-diyl))diethanone; MEK inhibitor I

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 'GH21+PD-1'Group (Experimental): GH21 combined with previous PD-1.
  Interventions: Drug: PD-1; Drug: GH21
- 'GH21+ALK Inhibitor'Group (Experimental): GH21 combined with previous ALK inhibitor.
  Interventions: Drug: ALK inhibitor; Drug: GH21
- 'GH21+MET Inhibitor'Group (Experimental): GH21 combined with previous MET inhibitor.
  Interventions: Drug: MET inhibitor; Drug: GH21
- 'GH21+BRAF Inhibitor+MEK Inhibitor'Group (Experimental): GH21 combined with previous BRAF inhibitor and MEK inhibitor.
  Interventions: Drug: BRAF Inhibito; Drug: GH21; Drug: MEK Inhibitor
- 'GH21+EGFR Monoclonal Antibody'Group (Experimental): GH21 combined with previous EGFR Monoclonal Antibody.
  Interventions: Drug: EGFR Monoclonal antibody; Drug: GH21

INTERVENTIONS:
Drug: PD-1 — Previous PD-1
  Arms: 'GH21+PD-1'Group
Drug: MET inhibitor — Previous MET inhibitor
  Arms: 'GH21+MET Inhibitor'Group
Drug: ALK inhibitor — Previous ALK inhibitor
  Arms: 'GH21+ALK Inhibitor'Group
Drug: BRAF Inhibito — Previous BRAF inhibitor
  Arms: 'GH21+BRAF Inhibitor+MEK Inhibitor'Group
Drug: EGFR Monoclonal antibody — Previous EGFR Monoclonal antibody
  Arms: 'GH21+EGFR Monoclonal Antibody'Group
Drug: GH21 — Oral, 15mg BIW or 6mg QD
Drug: MEK Inhibitor — Previous MEK Inhibitor
  Arms: 'GH21+BRAF Inhibitor+MEK Inhibitor'Group

SUMMARY:
This study is aim to evaluate the preliminary efficacy of GH21 combined with previous target therapy or immunotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study preset two dose groups, dose group 1 is GH21 15 mg (BIW, D1D2) combined with ALK inhibitor, or MET inhibitor, or BRAF inhibitor +MEK inhibitor, or PD-1 inhibitor, or EGFR monoantibody, or other drugs such as FGFR inhibitor, and it is planned to enroll up to 36 subjects. Dose group 2 was GH21 6 mg (QD) combined with ALK inhibitor, or MET inhibitor, or BRAF inhibitor +MEK inhibitor, or PD-1 inhibitor, or EGFR monoclonal antibody, or other drugs such as FGFR inhibitor, and was planned to enroll up to 36 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their legal representatives can understand and voluntarily sign the written ICF (before the start of screening and any study procedures);
2. Male or female subjects aged ≥18 years;
3. Patients with advanced solid tumors confirmed by cytological or histological assessments;
4. Patients have at least one measurable lesion as defined by RECIST v1.1 (a tumor lesion in the area that has undergone radiotherapy or other loco-regional therapies, is generally not considered as measurable unless there is a disease progression in the lesion);
5. Life expectancy of ≥ 3 months;
6. ECOG PS score of 0-1;
7. The subjects must have adequate organ functions;
8. Male and female of reproductive potential must agree to take reliable contraceptive measures (hormone or barrier methods or abstinence) from signing the ICF until 6 months after the last dose. Pregnancy test results must be negative for female of reproductive potential within 7 days prior to the first dose of the investigational product.

Exclusion Criteria:

1. Subjects who receive any chemotherapy or antitumor biologics within 3 weeks, or antitumor therapies such as radiotherapy and endocrine therapy within 4 weeks prior to the first dose of the investigational product, except for the following:

   * Use of nitrosoureas or mitomycin C within 6 weeks prior to the first dose of the investigational product;
   * Oral administration of fluorouracils, small molecule targeted drugs, and Chinese herbal medicines or Chinese patent medicines with antitumor indications within 5 half-lives or 2 weeks before the first dose of the investigational product (whichever is shorter);
   * Small molecule TKI inhibitors within 5 half-lives or 2 weeks prior to the first dose of the investigational product (whichever is shorter);
   * Local palliative radiotherapy within 2 weeks prior to the first dose of the investigational product; Note: If the latest anti-tumor therapy before enrollment is only the intended combination therapy, follow-up therapy can be carried out according to the original treatment cycle according to clinical needs, without waiting for elution.
2. Subjects who have had another investigational new drug or therapy within 4 weeks prior to the first dose of the investigational product;
3. Subjects who have had a major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose of the investigational product, or require an elective surgery during the study;
4. Subjects who have received strong P-gp inhibitors or inducers within 2 weeks or within 5 half-lives prior to the first dose of the investigational product;
5. Subjects with evidence of the following heart conditions:

   * Acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, cerebrovascular accident, or transient ischemic attack within 6 months prior to the first dose of the investigational product;
   * Grade III-IV heart failure diagnosed according to the cardiac function classification of the New York Heart Association at screening;
   * Echocardiography (ECHO) shows the left ventricular ejection fraction (LVEF) ≤ 50% at screening;
   * QT interval corrected by Fridericia method (QTcF) is ≥ 450 ms (male) or ≥ 470 ms (female) at screening;
   * Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) despite of medication treatment at screening;
6. Subjects with dysphagia, gastrointestinal disorders that affect drug absorption, or other malabsorption conditions, such as intestinal obstruction, Crohn's disease, ulcerative colitis, short bowel syndrome, delayed gastric emptying, or severe gastrointestinal toxicities that have not resolved to Grade 2 or lower prior to the first dose of the investigational product; or subjects are diagnosed with a clinically significant or acute gastrointestinal disease;
7. Subjects with Uncontrolled pleural effusion, pericardial effusion, or pleural effusion requiring repeated drainage (once a month or more frequently);
8. Subjects with active central nervous system metastasis and/or carcinomatous meningitis (e.g., brain metastases accompanied by central nervous system symptoms, including headache, vomiting and dizziness, etc.);
9. Subjects with interstitial pneumonia, or any evidence of clinically active interstitial lung disease within 6 months before the first dose of the investigational product;
10. Sujects with arteriovenous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks), venous thrombosis, and pulmonary embolism, occurred within 6 months before the first dose of the investigational product;
11. Subjects with a history of other malignancies (excluding those deemed eligible by the investigator, such as skin squamous cell carcinoma in situ, basal cell carcinoma, and cervical cancer in situ that have been cured and have not relapsed for 5 years);
12. Subjects with a history of severe allergies, a history of allergies to the investigational drug/any excipient/combination drug, or to multiple drugs;
13. Subjects with hepatitis B virus infection (HBsAg positivity and DNA copies < 100 IU/mL); or hepatitis C virus infection (HCV antibody positivity, and HCV RNA > ULN); or human immunodeficiency virus infection (HIV antibody positivity); or infected with treponema pallidum (defined as TP-Ab positive);
14. Subjects with active infections requiring anti-infective treatment (Grade ≥ 2) or fever > 38°C of unknown etiology within 28 days prior to the first dose of the investigational product;
15. Subjects with autoimmune diseases in the active phase within 28 days prior to the first dose of the investigational product;
16. Subjects with any toxicity caused by a previous antitumor therapy that has not resolved to Grade ≤ 1 according to CTCAE 5.0 (except for alopecia, Grade 2 peripheral neuropathy, and/or other Grade ≤ 2 AEs of insignificant safety risks) before the first dose of the investigational product;
17. Female subjects who are pregnant or breastfeeding;
18. Subjects who are not suitable for this study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Based on RECIST 1.1 Criteria | 3 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 3 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments.
Duration of Response (DOR) Based on RECIST 1.1 Criteria | 3 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy termination, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR）Based on RECIST 1.1 Criteria | 3 years
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD).
Progression-Free Survival (PFS) Based on RECIST 1.1 Criteria | 3 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.
Plasma Peak Concentration (Cmax) | 3 years
  Highest observed plasma concentration of GH21.
Time to Achieve Cmax (Tmax) | 3 years
  Time of highest observed plasma concentration of GH21.
Area under the Plasma Concentration-Time Curve (AUC) | 3 years
  Area under the plasma concentration-time curve of GH21.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Doctorate, Principal Investigator — +86-10-87788495; Haidan Wang, Doctorate, Study Director — +86-512-86861608
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu